CLINICAL TRIAL: NCT03167203
Title: A Safety Surveillance Study of Events of Special Interest Occurring in Subjects With Macular Degenerative Disease Treated With Human Embryonic Stem Cell-derived Retinal Pigment Epithelial Cell Therapy
Brief Title: A Safety Surveillance Study in Subjects With Macular Degenerative Disease Treated With Human Embryonic Stem Cell-derived Retinal Pigment Epithelial Cell Therapy
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Institute for Regenerative Medicine (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7316-CL-0007; 2016-005245-23 (EudraCT Number); RPE-SSS-001 (Other: Sponsor)
Record Dates: First submitted 2017-05-24; First posted 2017-05-25 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Macular Degenerative Disease
Keywords: hESC-RPE; Macular Degenerative Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- hESC-RPE cells (Experimental): Participants previously enrolled into an Astellas Institute for Regenerative Medicine (AIRM) sponsored clinical trial and treated with Human Embryonic Stem Cell-Derived Retinal Pigment Epithelial (hESC-RPE) cells
  Interventions: Biological: Human Embryonic Stem Cell-Derived Retinal Pigment Epithelial Cells

INTERVENTIONS:
Biological: Human Embryonic Stem Cell-Derived Retinal Pigment Epithelial Cells — Participants who have received sub-retinal transplant of hESC-RPE cells in an AIRM sponsored clinical trial
  Other Names: ASP7316

SUMMARY:
The purpose of this study is to is to evaluate the occurrence of late onset (i.e., greater than 5 years after treatment) adverse events of special interest (AESI) in participants who have received sub-retinal transplant of human embryonic stem cell derived - retinal pigment epithelial (hESC-RPE) cells in an AIRM-sponsored clinical trial. The events of special interest are adverse events (AEs) that are presumed to have a potential causal relationship to the hESC-RPE cells.

DETAILED DESCRIPTION:
Participants will be contacted by the Patient Outreach Center (POC) on an annual basis to complete a questionnaire about the occurrence of AESI, as defined in the Outcome Measure section.

The questionnaire will be completed directly by the participant (via a secure web based platform) or will be administered via telephone by a POC staff member. In the event of the occurrence of a AESI, study participant will be encouraged to contact the POC as soon as possible, rather than wait for the annual questionnaire completion. Follow up data is inclusive of the 1 year in the core trial, 4 years in the long term follow up trial and 10 years in this long term safety follow up. Participation for United Kingdom participants will be life-long.

ELIGIBILITY:
Inclusion Criteria:

* Participant was treated with hESC-RPE cell therapy in an Astellas Institute for Regenerative Medicine (AIRM) sponsored clinical trial in macular degenerative disease.
* Participant is able to understand.

Exclusion Criteria:

* There are no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events (AEs) that are ophthalmologic, neurologic, infectious or hematologic | Up to 15 Years
  Adverse events (AEs) will be coded using Medical Dictionary for Regulatory Activities (MedDRA). Participant self-reported via an annual questionnaire of adverse events that are ophthalmologic, neurologic, infectious or hematologic.
Number of new diagnoses of an immune-mediated disorder | Up to 15 Years
  Any new diagnosis of an immune-mediated disorder will be participant self-reported via an annual questionnaire.
Incidents of new cancer, irrespective of prior history | Up to 15 Years
  Any new cancer, irrespective of prior history, will be participant self-reported via an annual questionnaire.
Incidents of hESC-RPE cell proliferation | Up to 15 Years
  Occurrence of human embryonic stem cell derived - retinal pigment epithelial (hESC-RPE) cell proliferation will be participant self-reported via an annual questionnaire.
Incidents of ectopic tissue (RPE or non-RPE) formation | Up to 15 Years
  Occurrence of ectopic tissue (retinal pigment epithelial [RPE] or non-RPE) will be participant self-reported via an annual questionnaire
Number of participant reported pregnancies or pregnancy of participant's partner | Up to 15 Years
  Occurrence of pregnancy will be participant self-reported via an annual questionnaire
Number of reported pregnancy outcome(s) | Up to 15 Years
  Occurrence of pregnancy outcomes will be participant self-reported via an annual questionnaire
All cause death | Up to 15 Years
  All causes of death will be collected via an annual questionnaire (through participant-designated secondary contacts)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Institute for Regenerative Medicine
Locations (2):
- Private Practice, Kansas City, Missouri, United States
- Site GB44001, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/